CLINICAL TRIAL: NCT05746455
Title: Motivation Skills Training to Enhance Functional Outcomes for People With Schizophrenia (Open Trial)
Brief Title: Motivation Skills Training for Schizophrenia
Acronym: MST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alice Saperstein, PhD, Associate Professor of Medical Psychology (in Psychiatry), Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8394-1; 1R34MH129552-01A1 (NIH)
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Motivation; Skills Training
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Open Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivation Skills Training (MST) (Experimental): Participants will complete a baseline assessment, receive weekly MST sessions in a group format for a duration of 12 weeks, and will then repeat the assessment battery from baseline as well as a satisfaction survey.
  Interventions: Behavioral: Motivation Skills Training (MST)

INTERVENTIONS:
Behavioral: Motivation Skills Training (MST) — MST is a weekly group-based skills training intervention that aims to improve knowledge about one's level and sources of motivation, the ability to monitor and regulate (understand and manage) motivation, so that one can better initiate and sustain goal-directed behavior.

SUMMARY:
This study will take place at one outpatient clinic serving adults with serious mental illness and will recruit ten individuals (N=10) with a DSM-5 diagnosis of schizophrenia or schizoaffective disorder to participate in an Open Trial of Motivation Skills Training (MST). MST is a weekly group-based skills training intervention that aims to improve knowledge about one's level and sources of motivation, the ability to monitor and regulate (understand and manage) motivation, so that one can better initiate and sustain goal-directed behavior. Participants who consent for research will complete assessments of motivation, goal attainment, quality of life, executive functioning, community functioning, and psychiatric symptoms severity. The intervention phase will be approximately 12 weeks in duration and will entail weekly MST group sessions. At treatment endpoint, participants will be asked to repeat the assessment battery from baseline as well as a satisfaction survey. Change in motivation, goal attainment and quality of life will indicate whether MST is engaging the hypothesized target (motivation) and whether there is impact on functioning.

DETAILED DESCRIPTION:
Schizophrenia is a major public health problem associated with core motivational deficits that are amongst the strongest predictors of impaired functional outcomes. Without motivation, people are unable to maintain their pursuit of employment or educational goals, engage in treatment, and regularly participate in healthy life decisions. Current pharmacological and psychosocial treatments for schizophrenia have demonstrated limited effectiveness for improving this core symptom. Motivation Skills Training (MST) is a novel intervention that addresses this clinical need. The premise of MST is that knowledge about one's level and sources of motivation underlies the ability to regulate (i.e., understand and manage) motivation, and that motivation self-regulation can in turn facilitate task initiation and persistence. By facilitating goal-directed behavior, MST aims to enhance daily functioning and goal attainment in people with schizophrenia. MST teaches people about motivation and how to self-regulate motivation, empowering individuals to become active agents in controlling their own motivation and behavior. This study uses a 2-phase model of intervention testing to establish the feasibility, acceptability and pilot effectiveness of MST for adults ages 18-65 with a schizophrenia spectrum diagnosis. An initial open trial of MST in one outpatient clinic will provide stakeholder input on the acceptability and clinical utility of MST content and format, informing refinements to the treatment manual. A subsequent randomized controlled trial will test the effectiveness of MST versus a Healthy Behaviors Control (HBC) group, both conducted in the context of routine recovery-oriented services.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. A primary Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnosis of schizophrenia or schizoaffective disorder
3. Medically and psychiatrically stable outpatient status
4. English Fluency

Exclusion Criteria:

1. Indications of Intellectual Disability as documented in medical history or measured by < 70 premorbid full scale Intelligence Quotient (IQ) estimate
2. Severe substance use within the past 3 months determined by DSM-5 criteria
3. Neurologic condition causing brain disease
4. Mild to severe cognitive impairment associated with possible dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Saperstein, PhD, Principal Investigator — Columbia University
Locations (1):
- The Bridge Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be made available to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with public repositories such as the National Institute of Mental Health (NIMH) Data Archive. Data will include demographic information, baseline and post raw data derived from primary and secondary outcome measures.
Time Frame: A list of all data expected will be submitted by July 10, 2023. Subsequently raw data will be submitted on a semi-annual basis. Unpublished de-identified data will be submitted prior to study completion and will be shared within one year after project completion or when the data are published, whichever is earlier.
Access Criteria: Data in NIH repositories may be accessed through the NIH Data Access Committee which reviews data access and submission requests.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivation Skills Training (MST)
Started | 8 (Started indicates participants (N) who completed baseline assessments of motivation, goals, and quality of life)
Completed | 6 (Completed indicates participants (N) who completed post-treatment assessments of motivation, goals, and quality of life.)
Not Completed | 2
Not completed — Discharged from Clinical Service | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Motivation Skills Training (MST)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.375 (12.489)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 1
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Motivation and Pleasure (MAP) Scale [Mean (Standard Deviation); unit: score on a scale] | 2.39 (0.60)

OUTCOME MEASURES:

1. Primary Outcome: Change in Motivation and Pleasure Scale (MAP)
Description: MAP is an interviewer rated measure of motivation, pleasure, and engagement in work, school, recreational and social activities. Possible total scores range from 0 to 36, with lower scores indicating better outcomes. The average MAP score ranges from 0-4 with lower scores indicating better outcomes.
Time Frame: Baseline and up to 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivation Skills Training (MST)
Number analyzed (Participants) | 6
score on a scale | 0.50 (0.33)

2. Primary Outcome: Change in Goal Attainment Scaling (GAS)
Description: GAS measures progress towards personal goal attainment, rated along a continuum of predetermined successful outcomes on a scale from 0 to 10. Higher scores indicate better outcomes.
Time Frame: Baseline and up to 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivation Skills Training (MST)
Number analyzed (Participants) | 6
score on a scale | 2.0 (1.2)

3. Secondary Outcome: Change in Heinrichs Carpenter Quality of Life Scale (QLS)
Description: QLS is a semi-structured interview which evaluates psychosocial functional outcome. QLS is scored by summing the 7 items reflecting four domains: interpersonal functioning, intrapsychic foundations, instrumental role function, and common objects/activities. Total scores ranges from 0 to 42 where higher scores indicate better functioning.
Time Frame: Baseline and up to 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivation Skills Training (MST)
Number analyzed (Participants) | 6
score on a scale | 5.17 (2.92)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for 4 months inclusive of the dates from study start to completion.
Arm/Group | Motivation Skills Training (MST)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT05746455/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT05746455/SAP_001.pdf